CLINICAL TRIAL: NCT02388529
Title: A Randomized, Double-Blinded, Placebo-Controlled, Multiple Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics and Efficacy of Bendavia™ (MTP-131) in Patients With Heart Failure Due to Reduced Left Ventricular Ejection Fraction
Brief Title: A Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of Bendavia™ (MTP-131) in Patients With Heart Failure
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPIHF-202
Record Dates: First submitted 2015-03-01; First posted 2015-03-17 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure
Keywords: Heart Failure; Bendavia™; MTP-131
MeSH Terms: conditions — Heart Failure | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose (Experimental)
  Interventions: Drug: MTP-131
- Intermediate dose (Experimental)
  Interventions: Drug: MTP-131
- High dose (Experimental)
  Interventions: Drug: MTP-131
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MTP-131 — MTP-131 (low dose) administered as once-daily 1- hour intravenous infusion for 5 consecutive days
  Arms: Low dose
Drug: MTP-131 — MTP-131 (intermediate dose) administered as once-daily 1- hour intravenous infusion for 5 consecutive days
  Arms: Intermediate dose
Drug: MTP-131 — MTP-131 (high dose) administered as once-daily 1- hour intravenous infusion for 5 consecutive days
  Arms: High dose
Drug: Placebo — Placebo Comparator (at each dose cohort) administered as once-daily 1- hour intravenous infusion for 5 consecutive days
  Arms: Placebo

SUMMARY:
This study is a single-center, randomized, double-blind, placebo-controlled study in patients with stable heart failure to evaluate the safety, tolerability, pharmacokinetics, and efficacy of multiple ascending doses of Bendavia™ (MTP-131) intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

* LVEF ≤45% by 2-D echocardiogram.
* Diagnosis of New York Heart Association Class II or III HF for a minimum of 6 months prior to the Screening Visit.
* HF is considered to be stable, in the judgment of the Principal Investigator and no hospitalization related to HF has occurred within the 1 month prior to the Screening Visit.
* Treatment with appropriate pharmacologic therapy for HF including, but not limited to, angiotensin converting enzyme inhibitor (ACEI) and/or angiotensin receptor blocker (ARB), and an evidence-based beta blocker for the treatment of HF
* Females of child-bearing potential must have a negative serum pregnancy test at the Screening Visit.
* Written informed consent obtained that strictly adheres to the written guidelines from the local Ethical Committee (EC).

Exclusion Criteria:

* Unstable angina pectoris within 1 month before initiation of screening procedures. Unstable angina is defined as the occurrence of chest pain more frequently than usual, pain at rest or upon minimal exertion, or protracted episodes of pain without any discernible trigger, and/or chest pain that persists despite use of vasodilatory therapy (e.g., nitroglycerin).
* Coronary or peripheral artery revascularization procedure within 2 months prior to the Screening Visit.
* An acute myocardial infarction within 3 months prior to the Screening Visit.
* Supine resting heart rate ≥ 100 beats per minute after 5 minutes rest.
* Uncontrolled hypertension defined as a systolic blood pressure (BP) >180 mm Hg or a diastolic BP >110 mm Hg on at least 2 consecutive readings.
* Requirement for valve or other cardiac surgery (e.g., pericardectomy).
* Cardiac surgery or valvuloplasty within 2 month prior to the Screening Visit.
* General surgery within 1 month prior to the Screening Visit.
* Restrictive cardiomyopathy, obstructive cardiomyopathy, pericardial disease, amyloidosis, infiltrative cardiomyopathy, uncorrected thyroid disease, or dyskinetic left ventricular aneurysm.
* Cerebrovascular accident or transient ischemic attack within 3 months prior to the Screening Visit.
* Liver enzyme (alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST]) elevation >3x the upper limit of normal (ULN).
* Estimated glomerular filtration rate (eGFR) <30 mL/min, using the Modification of Diet in Renal Disease (MDRD) Study equation.
* Known active drug or alcohol abuse.
* Active infection requiring systemic treatment or surgical intervention.
* Significant acute or chronic medical or psychiatric illness that, in the judgment of the Investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study.
* Female patients who are pregnant or breastfeeding.

  * Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Assessed up to Day 33
Mean peak plasma concentration (Cmax) of MTP-131 (ng/ml) in each cohort | Assessed up to Day 12

SECONDARY OUTCOMES:
Changes in echocardiographic LV end-systolic volume (LVESV) | Assessed up to Day 33

CONTACTS AND LOCATIONS:
Overall Officials: Jim Carr, PharmD, Study Director — Stealth BioTherapeutics Inc.; Sotir Marchev, MD,PhD, FESC, Principal Investigator — Bulgaria
Locations (1):
- Sevlievo, Gabrovo, Bulgaria